CLINICAL TRIAL: NCT06417034
Title: Hand Training Device For Cognitive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: A-ER-110-485
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Healthy Elderly; Mild Cognitive Impairment (MCI)
Keywords: Functional near infrared spectroscopy; Parameters of digit force independence; Pressing Evaluation and Training System
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-based game training (Experimental): Subjects will be asked to press their finger while a series of archery target continuously drop down and pass by the bottom line follow the beats of music melody on Tipr.
  Interventions: Device: Game Software
- Non music-based game training (Active Comparator): The background music will be disabled. Subjects need to press equally amount of force in certain tolerance that been set by only the visual cue on Tipr.
  Interventions: Device: Game Software

INTERVENTIONS:
Device: Game Software — The software is interfaced with a modified version of Frets on Fire (FOF)-an open source computer game similar to Guitar Hero.

SUMMARY:
Previous studies indicated that auditory stimulation as an external cue might have positive impacts on sensorimotor synchronization. Additionally, according to previous reports apart from traditional interventions, digitized game-based device, such as FTOMBVG, are beneficial for the brain activation in elderly. Moreover, enhanced finger force control and coordination lead to better hand dexterity and is believed to eventually improve life independence in the healthy elderly and the elderly with cognitive decline. Therefore, this study aims to develop an advanced systems based on the previous one, that can provide hand function rehabilitation, cognitive training, and emotional comfort for the elderly or people suffer from cognitive deficiency. They can enhance their finger force control or visual to motor synchronization by music embedded during the gaming process.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate in Mandarin Chinese or Taiwanese
* MCI, according to clinical neurological assessment, Montreal Cognitive Assessment (MoCA):≦25&≧19
* Ability to perform ADL independently, no hand function disability
* Voluntarily participation and ability to sign the informed consent form

Exclusion Criteria:

* Alzheimers disease diagnosed by physicians or meeting the diagnostic criteria for dementia
* Physician's diagnosis of stroke
* Any mental illness or behavior problems and inability to cooperate with the trainer
* Visual impairment or hand diseases resulting in an inability to perform finger press
* received other cognitive or physical training in the past year
* any sight, hearing, or communication impairment

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) | 30 minutes
  The Oxygenated hemoglobin (HbO) was measured while the participants play the game under both conditions
Montreal Cognitive Assessment (MoCA) test | 10 minutes
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: Short term memory, Visuospatial abilities, Executive functions, Attention, concentration and working memory, Language, Orientation to time and place. The sensitivity of MoCA for detecting MCI is 90%.
EN value | 5 minutes
  The force independence is collected from the data during force control game in each evaluation session. The parameter of force independence is an index of five digits overall enslaving presented as EN.

SECONDARY OUTCOMES:
Maximum voluntary isometric contraction (MVIC) | 10 seconds
  Maximum voluntary isometric contraction of each digit is measured for training reference.

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, PhD, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Organization, W.H., Global health and aging. Geneva: World Health Organization, 2011.
- [Background] Olshansky SJ, Ault AB. The fourth stage of the epidemiologic transition: the age of delayed degenerative diseases. Milbank Q. 1986;64(3):355-91. PMID 3762504
- [Background] Sun Y, Lee HJ, Yang SC, Chen TF, Lin KN, Lin CC, Wang PN, Tang LY, Chiu MJ. A nationwide survey of mild cognitive impairment and dementia, including very mild dementia, in Taiwan. PLoS One. 2014 Jun 18;9(6):e100303. doi: 10.1371/journal.pone.0100303. eCollection 2014. PMID 24940604
- [Background] Wimo A, Guerchet M, Ali GC, Wu YT, Prina AM, Winblad B, Jonsson L, Liu Z, Prince M. The worldwide costs of dementia 2015 and comparisons with 2010. Alzheimers Dement. 2017 Jan;13(1):1-7. doi: 10.1016/j.jalz.2016.07.150. Epub 2016 Aug 29. PMID 27583652
- [Background] Langa KM, Levine DA. The diagnosis and management of mild cognitive impairment: a clinical review. JAMA. 2014 Dec 17;312(23):2551-61. doi: 10.1001/jama.2014.13806. PMID 25514304
- [Background] Maioli F, Coveri M, Pagni P, Chiandetti C, Marchetti C, Ciarrocchi R, Ruggero C, Nativio V, Onesti A, D'Anastasio C, Pedone V. Conversion of mild cognitive impairment to dementia in elderly subjects: a preliminary study in a memory and cognitive disorder unit. Arch Gerontol Geriatr. 2007;44 Suppl 1:233-41. doi: 10.1016/j.archger.2007.01.032. PMID 17317458
- [Background] Abou Kassm S, Naja W, Hoertel N, Limosin F. [Pharmacological management of delusions associated with dementia]. Geriatr Psychol Neuropsychiatr Vieil. 2019 Sep 1;17(3):317-326. doi: 10.1684/pnv.2019.0813. French. PMID 31449050
- [Background] Folch J, Busquets O, Ettcheto M, Sanchez-Lopez E, Castro-Torres RD, Verdaguer E, Garcia ML, Olloquequi J, Casadesus G, Beas-Zarate C, Pelegri C, Vilaplana J, Auladell C, Camins A. Memantine for the Treatment of Dementia: A Review on its Current and Future Applications. J Alzheimers Dis. 2018;62(3):1223-1240. doi: 10.3233/JAD-170672. PMID 29254093
- [Background] Groot C, Hooghiemstra AM, Raijmakers PG, van Berckel BN, Scheltens P, Scherder EJ, van der Flier WM, Ossenkoppele R. The effect of physical activity on cognitive function in patients with dementia: A meta-analysis of randomized control trials. Ageing Res Rev. 2016 Jan;25:13-23. doi: 10.1016/j.arr.2015.11.005. Epub 2015 Nov 28. PMID 26607411
- [Background] Brasure M, Desai P, Davila H, Nelson VA, Calvert C, Jutkowitz E, Butler M, Fink HA, Ratner E, Hemmy LS, McCarten JR, Barclay TR, Kane RL. Physical Activity Interventions in Preventing Cognitive Decline and Alzheimer-Type Dementia: A Systematic Review. Ann Intern Med. 2018 Jan 2;168(1):30-38. doi: 10.7326/M17-1528. Epub 2017 Dec 19. PMID 29255839
- [Background] Baird A, Samson S. Music and dementia. Prog Brain Res. 2015;217:207-35. doi: 10.1016/bs.pbr.2014.11.028. Epub 2015 Jan 31. PMID 25725917
- [Background] Woods B, O'Philbin L, Farrell EM, Spector AE, Orrell M. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2018 Mar 1;3(3):CD001120. doi: 10.1002/14651858.CD001120.pub3. PMID 29493789
- [Background] Spector A, Orrell M, Woods B. Cognitive Stimulation Therapy (CST): effects on different areas of cognitive function for people with dementia. Int J Geriatr Psychiatry. 2010 Dec;25(12):1253-8. doi: 10.1002/gps.2464. PMID 20069533
- [Background] Spector A, Orrell M, Davies S, Woods B. Reality orientation for dementia. Cochrane Database Syst Rev. 2000;(4):CD001119. doi: 10.1002/14651858.CD001119. PMID 11034699
- [Background] Diaz-Perez E, Florez-Lozano JA. [Virtual reality and dementia]. Rev Neurol. 2018 May 16;66(10):344-352. Spanish. PMID 29749595
- [Background] Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. Ageing Res Rev. 2013 Jan;12(1):263-75. doi: 10.1016/j.arr.2012.07.003. Epub 2012 Jul 25. PMID 22841936
- [Background] Lam NW, Goh HT, Kamaruzzaman SB, Chin AV, Poi PJ, Tan MP. Normative data for hand grip strength and key pinch strength, stratified by age and gender for a multiethnic Asian population. Singapore Med J. 2016 Oct;57(10):578-584. doi: 10.11622/smedj.2015164. Epub 2015 Nov 13. PMID 26768064
- [Background] Y. Fu, D.-H. Wang, Cognitive aging and the brain: HAROLD model debate, Adv. Psychol. Sci. 17 86- 91 (2009).
- [Background] Scherder E, Dekker W, Eggermont L. Higher-level hand motor function in aging and (preclinical) dementia: its relationship with (instrumental) activities of daily life--a mini-review. Gerontology. 2008;54(6):333-41. doi: 10.1159/000168203. Epub 2008 Nov 11. PMID 18997468
- [Background] Volkers KM, Scherder EJ. Physical performance is associated with working memory in older people with mild to severe cognitive impairment. Biomed Res Int. 2014;2014:762986. doi: 10.1155/2014/762986. Epub 2014 Mar 16. PMID 24757674
- [Background] Fauth EB, Schaefer SY, Zarit SH, Ernsth-Bravell M, Johansson B. Associations Between Fine Motor Performance in Activities of Daily Living and Cognitive Ability in a Nondemented Sample of Older Adults: Implications for Geriatric Physical Rehabilitation. J Aging Health. 2017 Oct;29(7):1144-1159. doi: 10.1177/0898264316654674. Epub 2016 Jun 22. PMID 27339106
- [Background] Babiloni C, Frisoni GB, Pievani M, Vecchio F, Infarinato F, Geroldi C, Salinari S, Ferri R, Fracassi C, Eusebi F, Rossini PM. White matter vascular lesions are related to parietal-to-frontal coupling of EEG rhythms in mild cognitive impairment. Hum Brain Mapp. 2008 Dec;29(12):1355-67. doi: 10.1002/hbm.20467. PMID 17979121
- [Background] Imran MB, Kawashima R, Awata S, Sato K, Kinomura S, Ono S, Sato M, Fukuda H. Tc-99m HMPAO SPECT in the evaluation of Alzheimer's disease: correlation between neuropsychiatric evaluation and CBF images. J Neurol Neurosurg Psychiatry. 1999 Feb;66(2):228-32. doi: 10.1136/jnnp.66.2.228. PMID 10071106
- [Background] Ehrsson HH, Fagergren E, Forssberg H. Differential fronto-parietal activation depending on force used in a precision grip task: an fMRI study. J Neurophysiol. 2001 Jun;85(6):2613-23. doi: 10.1152/jn.2001.85.6.2613. PMID 11387405
- [Background] Umetsu A, Okuda J, Fujii T, Tsukiura T, Nagasaka T, Yanagawa I, Sugiura M, Inoue K, Kawashima R, Suzuki K, Tabuchi M, Murata T, Mugikura S, Higano S, Takahashi S, Fukuda H, Yamadori A. Brain activation during the fist-edge-palm test: a functional MRI study. Neuroimage. 2002 Sep;17(1):385-92. doi: 10.1006/nimg.2002.1218. PMID 12482091
- [Background] Sawamoto N, Honda M, Hanakawa T, Aso T, Inoue M, Toyoda H, Ishizu K, Fukuyama H, Shibasaki H. Cognitive slowing in Parkinson disease is accompanied by hypofunctioning of the striatum. Neurology. 2007 Mar 27;68(13):1062-8. doi: 10.1212/01.wnl.0000257821.28992.db. PMID 17389313
- [Background] Zhang N, Yuan X, Li Q, Wang Z, Gu X, Zang J, Ge R, Liu H, Fan Z, Bu L. The effects of age on brain cortical activation and functional connectivity during video game-based finger-to-thumb opposition movement: A functional near-infrared spectroscopy study. Neurosci Lett. 2021 Feb 16;746:135668. doi: 10.1016/j.neulet.2021.135668. Epub 2021 Jan 23. PMID 33497717
- [Background] Chen LL, Li H, Chen XH, Jin S, Chen QH, Chen MR, Li N. Effects of Hand Exercise on Eating Action in Patients With Alzheimer's Disease. Am J Alzheimers Dis Other Demen. 2019 Feb;34(1):57-62. doi: 10.1177/1533317518803722. Epub 2018 Oct 9. PMID 30301358
- [Background] de Boer C, Echlin HV, Rogojin A, Baltaretu BR, Sergio LE. Thinking-While-Moving Exercises May Improve Cognition in Elderly with Mild Cognitive Deficits: A Proof-of-Principle Study. Dement Geriatr Cogn Dis Extra. 2018 Jul 11;8(2):248-258. doi: 10.1159/000490173. eCollection 2018 May-Aug. PMID 30140274
- [Background] Gates NJ, Sachdev PS, Fiatarone Singh MA, Valenzuela M. Cognitive and memory training in adults at risk of dementia: a systematic review. BMC Geriatr. 2011 Sep 25;11:55. doi: 10.1186/1471-2318-11-55. PMID 21942932
- [Background] Sarkamo T, Ripolles P, Vepsalainen H, Autti T, Silvennoinen HM, Salli E, Laitinen S, Forsblom A, Soinila S, Rodriguez-Fornells A. Structural changes induced by daily music listening in the recovering brain after middle cerebral artery stroke: a voxel-based morphometry study. Front Hum Neurosci. 2014 Apr 17;8:245. doi: 10.3389/fnhum.2014.00245. eCollection 2014. PMID 24860466
- [Background] Bruscia KE. Defining Music Therapy. 3rd ed. University Park, IL: Barcelona Publishers; (2014).
- [Background] Wheeler BL. Music Therapy Handbook. New York: Guilford Publications; (2015).
- [Background] Robb SL, Hanson-Abromeit D, May L, Hernandez-Ruiz E, Allison M, Beloat A, Daugherty S, Kurtz R, Ott A, Oyedele OO, Polasik S, Rager A, Rifkin J, Wolf E. Reporting quality of music intervention research in healthcare: A systematic review. Complement Ther Med. 2018 Jun;38:24-41. doi: 10.1016/j.ctim.2018.02.008. Epub 2018 Mar 7. PMID 29857877
- [Background] Lim HB, Karageorghis CI, Romer LM, Bishop DT. Psychophysiological effects of synchronous versus asynchronous music during cycling. Med Sci Sports Exerc. 2014 Feb;46(2):407-13. doi: 10.1249/MSS.0b013e3182a6378c. PMID 24441216
- [Background] Ramji R, Aasa U, Paulin J, Madison G. Musical information increases physical performance for synchronous but not asynchronous running. Psychol Music.;44(5):984-95 (2016).
- [Background] Buhmann J, Moens B, Van Dyck E, Dotov D, Leman M. Optimizing beat synchronized running to music. PLoS One. 2018 Dec 6;13(12):e0208702. doi: 10.1371/journal.pone.0208702. eCollection 2018. PMID 30521634
- [Background] Jin X, Wang B, Lv Y, Lu Y, Chen J, Zhou C. Does dance training influence beat sensorimotor synchronization? Differences in finger-tapping sensorimotor synchronization between competitive ballroom dancers and nondancers. Exp Brain Res. 2019 Mar;237(3):743-753. doi: 10.1007/s00221-018-5410-4. Epub 2019 Jan 2. PMID 30600336
- [Background] Miura A, Kudo K, Ohtsuki T, Kanehisa H, Nakazawa K. Relationship between muscle cocontraction and proficiency in whole-body sensorimotor synchronization: a comparison study of street dancers and nondancers. Motor Control. 2013 Jan;17(1):18-33. doi: 10.1123/mcj.17.1.18. Epub 2012 Sep 7. PMID 22964842
- [Background] Friedman N, Chan V, Zondervan D, Bachman M, Reinkensmeyer DJ. MusicGlove: motivating and quantifying hand movement rehabilitation by using functional grips to play music. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:2359-63. doi: 10.1109/IEMBS.2011.6090659. PMID 22254815
- [Background] Han E, Park J, Kim H, Jo G, Do HK, Lee BI. Cognitive Intervention with Musical Stimuli Using Digital Devices on Mild Cognitive Impairment: A Pilot Study. Healthcare (Basel). 2020 Feb 25;8(1):45. doi: 10.3390/healthcare8010045. PMID 32106559
- [Background] Semjen A, Ivry RB. The coupled oscillator model of between-hand coordination in alternate-hand tapping: a reappraisal. J Exp Psychol Hum Percept Perform. 2001 Apr;27(2):251-65. doi: 10.1037//0096-1523.27.2.251. PMID 11318046
- [Background] Patel AD, Iversen JR, Chen Y, Repp BH. The influence of metricality and modality on synchronization with a beat. Exp Brain Res. 2005 May;163(2):226-38. doi: 10.1007/s00221-004-2159-8. Epub 2005 Jan 15. PMID 15654589
- [Background] Tierney A, Kraus N. The ability to move to a beat is linked to the consistency of neural responses to sound. J Neurosci. 2013 Sep 18;33(38):14981-8. doi: 10.1523/JNEUROSCI.0612-13.2013. PMID 24048827
- [Background] Blais M, Albaret JM, Tallet J. Is there a link between sensorimotor coordination and inter-manual coordination? Differential effects of auditory and/or visual rhythmic stimulations. Exp Brain Res. 2015 Nov;233(11):3261-9. doi: 10.1007/s00221-015-4394-6. Epub 2015 Aug 4. PMID 26238405
- [Background] Sarkamo T, Pihko E, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M, Tervaniemi M. Music and speech listening enhance the recovery of early sensory processing after stroke. J Cogn Neurosci. 2010 Dec;22(12):2716-27. doi: 10.1162/jocn.2009.21376. PMID 19925203
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Sarkamo T, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Pattern of Emotional Benefits Induced by Regular Singing and Music Listening in Dementia. J Am Geriatr Soc. 2016 Feb;64(2):439-40. doi: 10.1111/jgs.13963. No abstract available. PMID 26889849
- [Background] Sarkamo T, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Clinical and Demographic Factors Associated with the Cognitive and Emotional Efficacy of Regular Musical Activities in Dementia. J Alzheimers Dis. 2016;49(3):767-81. doi: 10.3233/JAD-150453. PMID 26519435
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Background] Pohl P, Dizdar N, Hallert E. The Ronnie Gardiner Rhythm and Music Method - a feasibility study in Parkinson's disease. Disabil Rehabil. 2013;35(26):2197-204. doi: 10.3109/09638288.2013.774060. Epub 2013 Mar 12. PMID 23480646
- [Background] Altenmuller E, Marco-Pallares J, Munte TF, Schneider S. Neural reorganization underlies improvement in stroke-induced motor dysfunction by music-supported therapy. Ann N Y Acad Sci. 2009 Jul;1169:395-405. doi: 10.1111/j.1749-6632.2009.04580.x. PMID 19673814
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Background] Jacobsen JH, Stelzer J, Fritz TH, Chetelat G, La Joie R, Turner R. Why musical memory can be preserved in advanced Alzheimer's disease. Brain. 2015 Aug;138(Pt 8):2438-50. doi: 10.1093/brain/awv135. Epub 2015 Jun 3. PMID 26041611
- [Background] Cotelli M, Manenti R, Brambilla M, Gobbi E, Ferrari C, Binetti G, Cappa SF. Cognitive telerehabilitation in mild cognitive impairment, Alzheimer's disease and frontotemporal dementia: A systematic review. J Telemed Telecare. 2019 Feb;25(2):67-79. doi: 10.1177/1357633X17740390. Epub 2017 Nov 8. PMID 29117794
- [Background] Burton RL, O'Connell ME. Telehealth Rehabilitation for Cognitive Impairment: Randomized Controlled Feasibility Trial. JMIR Res Protoc. 2018 Feb 8;7(2):e43. doi: 10.2196/resprot.9420. PMID 29422453
- [Background] Ty, J. et al. in Human Aspects of IT for the Aged Population. Social Media, Games and Assistive Environments. (eds Jia Zhou & Gavriel Salvendy) 575-587 (Springer International Publishing).
- [Background] Suzuki T, Shimada H, Makizako H, Doi T, Yoshida D, Tsutsumimoto K, Anan Y, Uemura K, Lee S, Park H. Effects of multicomponent exercise on cognitive function in older adults with amnestic mild cognitive impairment: a randomized controlled trial. BMC Neurol. 2012 Oct 31;12:128. doi: 10.1186/1471-2377-12-128. PMID 23113898
- [Background] Park S, Bak A, Kim S, Nam Y, Kim HS, Yoo DH, Moon M. Animal-Assisted and Pet-Robot Interventions for Ameliorating Behavioral and Psychological Symptoms of Dementia: A Systematic Review and Meta-Analysis. Biomedicines. 2020 Jun 2;8(6):150. doi: 10.3390/biomedicines8060150. PMID 32498454
- [Background] Bernabei V, De Ronchi D, La Ferla T, Moretti F, Tonelli L, Ferrari B, Forlani M, Atti AR. Animal-assisted interventions for elderly patients affected by dementia or psychiatric disorders: a review. J Psychiatr Res. 2013 Jun;47(6):762-73. doi: 10.1016/j.jpsychires.2012.12.014. Epub 2013 Jan 29. PMID 23369337
- [Background] Wu YH, Truglio TS, Zatsiorsky VM, Latash ML. Learning to combine high variability with high precision: lack of transfer to a different task. J Mot Behav. 2015;47(2):153-65. doi: 10.1080/00222895.2014.961892. Epub 2014 Nov 3. PMID 25365477
- [Background] Castilla D, Suso-Ribera C, Zaragoza I, Garcia-Palacios A, Botella C. Designing ICTs for Users with Mild Cognitive Impairment: A Usability Study. Int J Environ Res Public Health. 2020 Jul 17;17(14):5153. doi: 10.3390/ijerph17145153. PMID 32708861